CLINICAL TRIAL: NCT02278536
Title: Development of Non-invasive Prenatal Diagnostic Test for Multiple Gestation Pregnancies Based on Fetal DNA Isolated From Maternal Blood
Brief Title: Multiple Gestation Study
Status: Completed | Type: Observational
Sponsor: Natera, Inc. (Industry)
Collaborators: Houston Perinatal Associates (Unknown); Lyndhurst Clinical Research (Unknown); Dr. Carpenter Maternal Fetal Medicine Clinic (Unknown); San Diego Perinatal Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: 13-016-NPT
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Trisomy 13; Trisomy 18; Trisomy 21; Sex Chromosome Abnormalities
Keywords: Trisomy 13; Trisomy 18; Trisomy 21; Sex Chromosome Abnormalities; Monosomy X; XXX; XXY; XYY
MeSH Terms: conditions — Trisomy 13 Syndrome; Trisomy 18 Syndrome; Down Syndrome; Sex Chromosome Aberrations; Turner Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal and Paternal blood samples
  CVS or Amniocentesis sample (optional)
  Child saliva sample (optional)
  *Biospecimen retention is optional portion of consent form
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Multiple high risk gestation pregnancies: women pregnant with twins or triplets at high risk for aneuploidy
- Multiple low risk gestation pregnancies: women pregnant with twins or triplets at low risk for aneuploidy

SUMMARY:
The objectives of the clinical study are to demonstrate the accuracy of our new NATUS diagnostic method to determine the genetic health of the developing fetuses in a multiple gestation pregnancy from a maternal blood sample. The long term goal of this study will be the development of a method of minimally invasive prenatal diagnosis that has a higher sensitivity and lower false positive rate in the intended population (e.g. multiple gestation pregnancies) than any currently available screening tests. This will result in fewer unnecessary amniocenteses and CVS procedures, which are associated with a risk of miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older at enrollment
* Clinically confirmed multiple gestation pregnancy
* Gestational age between ≥ 9 weeks, 0 days and ≤26 weeks 0 days by best obstetrical estimate
* Able to provide informed consent

Exclusion Criteria:

* Women carrying singleton pregnancy
* Surrogate or egg donor used

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant Women
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2013-03; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be to confirm the diagnostic capability of NATUS risk results classified as positive result for aneuploidy, negative result for aneuploidy or 'no call.' | 2 years
  The chromosomal status will be determined from the CVS or amniocentesis results, if available. A cheek swab or saliva sample will be collected from live-born children if there are no CVS or amniocentesis results.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kirshon, MD, Principal Investigator — Houston Perinatal Associates; Robert Lamar Parker, MD, Principal Investigator — Lyndhurst Clinical Research; Robert Carpenter, MD, Principal Investigator — Office of Dr. Robert Carpenter; Zach Demko, PhD, Principal Investigator — Natera, Inc.
Locations (8):
- United States (6):
  - Natera, Inc., San Carlos, California
  - San Diego Perinatal Center, San Diego, California
  - Carnegie Hill Imaging for Women, New York, New York
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Office of Dr. Robert Carpenter, Houston, Texas
  - Houston Perinatal Associates, Houston, Texas
- Bangalore Fetal Medicine Centre, Bangalore, India
- Fetal Medicine & Gynaecology Centre, Petaling Jaya, Selangor, Malaysia

REFERENCES:
- [Background] Pergament E, Cuckle H, Zimmermann B, Banjevic M, Sigurjonsson S, Ryan A, Hall MP, Dodd M, Lacroute P, Stosic M, Chopra N, Hunkapiller N, Prosen DE, McAdoo S, Demko Z, Siddiqui A, Hill M, Rabinowitz M. Single-nucleotide polymorphism-based noninvasive prenatal screening in a high-risk and low-risk cohort. Obstet Gynecol. 2014 Aug;124(2 Pt 1):210-218. doi: 10.1097/AOG.0000000000000363. PMID 25004354
- [Background] Ehrich M, Deciu C, Zwiefelhofer T, Tynan JA, Cagasan L, Tim R, Lu V, McCullough R, McCarthy E, Nygren AO, Dean J, Tang L, Hutchison D, Lu T, Wang H, Angkachatchai V, Oeth P, Cantor CR, Bombard A, van den Boom D. Noninvasive detection of fetal trisomy 21 by sequencing of DNA in maternal blood: a study in a clinical setting. Am J Obstet Gynecol. 2011 Mar;204(3):205.e1-11. doi: 10.1016/j.ajog.2010.12.060. Epub 2011 Feb 18. PMID 21310373
- [Background] Palomaki GE, Kloza EM, Lambert-Messerlian GM, Haddow JE, Neveux LM, Ehrich M, van den Boom D, Bombard AT, Deciu C, Grody WW, Nelson SF, Canick JA. DNA sequencing of maternal plasma to detect Down syndrome: an international clinical validation study. Genet Med. 2011 Nov;13(11):913-20. doi: 10.1097/GIM.0b013e3182368a0e. PMID 22005709
- [Background] Sehnert AJ, Rhees B, Comstock D, de Feo E, Heilek G, Burke J, Rava RP. Optimal detection of fetal chromosomal abnormalities by massively parallel DNA sequencing of cell-free fetal DNA from maternal blood. Clin Chem. 2011 Jul;57(7):1042-9. doi: 10.1373/clinchem.2011.165910. Epub 2011 Apr 25. PMID 21519036
- [Background] Bianchi DW, Platt LD, Goldberg JD, Abuhamad AZ, Sehnert AJ, Rava RP; MatErnal BLood IS Source to Accurately diagnose fetal aneuploidy (MELISSA) Study Group. Genome-wide fetal aneuploidy detection by maternal plasma DNA sequencing. Obstet Gynecol. 2012 May;119(5):890-901. doi: 10.1097/AOG.0b013e31824fb482. PMID 22362253
- [Background] Palomaki GE, Deciu C, Kloza EM, Lambert-Messerlian GM, Haddow JE, Neveux LM, Ehrich M, van den Boom D, Bombard AT, Grody WW, Nelson SF, Canick JA. DNA sequencing of maternal plasma reliably identifies trisomy 18 and trisomy 13 as well as Down syndrome: an international collaborative study. Genet Med. 2012 Mar;14(3):296-305. doi: 10.1038/gim.2011.73. Epub 2012 Feb 2. PMID 22281937
- [Background] Norton ME, Brar H, Weiss J, Karimi A, Laurent LC, Caughey AB, Rodriguez MH, Williams J 3rd, Mitchell ME, Adair CD, Lee H, Jacobsson B, Tomlinson MW, Oepkes D, Hollemon D, Sparks AB, Oliphant A, Song K. Non-Invasive Chromosomal Evaluation (NICE) Study: results of a multicenter prospective cohort study for detection of fetal trisomy 21 and trisomy 18. Am J Obstet Gynecol. 2012 Aug;207(2):137.e1-8. doi: 10.1016/j.ajog.2012.05.021. Epub 2012 Jun 1. PMID 22742782
- [Background] Canick JA, Kloza EM, Lambert-Messerlian GM, Haddow JE, Ehrich M, van den Boom D, Bombard AT, Deciu C, Palomaki GE. DNA sequencing of maternal plasma to identify Down syndrome and other trisomies in multiple gestations. Prenat Diagn. 2012 Aug;32(8):730-4. doi: 10.1002/pd.3892. Epub 2012 May 14. PMID 22585317